CLINICAL TRIAL: NCT03732547
Title: A Phase II Study on the Safety and Therapeutic Effect of Combination of PolyIC and PD-1 mAb in Subjects With Unresectable Hepatocellular Carcinoma
Brief Title: Study of PolyIC and PD-1 mAb in Subjects With Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISLD-1
Record Dates: First submitted 2018-10-22; First posted 2018-11-06 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma; Polyinosinic-polycytidylic acid; PD-1 mAb
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Poly I-C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 'PolyIC plus PD-1 mAb' and 'PD-1 mAb' (Experimental): 'PolyIC plus PD-1 mAb' group: PolyIC, 2mg, i.m., every other day, for three weeks. PD-1 mAb, 200mg, i.v., every three weeks.
  'PD-1 mAb' group: PD-1 mAb, 200mg, i.v., every three weeks.
  Interventions: Drug: PD-1 mAb; Drug: PolyIC

INTERVENTIONS:
Drug: PD-1 mAb — Intravenous infusion of PD-1 mAb, 200mg, once a time, every three weeks.
  Other Names: Programmed cell death-1 monoclonal antibody
Drug: PolyIC — Intramuscular injection of polyIC, 2mg, every other day, for three weeks.
  Other Names: Polyinosinic-polycytidylic acid

SUMMARY:
When multi-kinase inhibitors based therapies (sorafenib and regorafenib) are limited in late-stage liver cancer patients, there is no alternative options. PD-1 blockade has became a promising immunotherapeutic strategy in many cancers. While it showed limited efficacy in liver cancer. Polyinosinic-polycytidylic acid (PolyIC) has been widely studied as a new anti-tumor drug and recent study showed that polyIC and PD-L1 mAb has a quite synergetic effect on the hepatocellular carcinoma (HCC). This study is aimed to evaluate the safety and efficacy of the combination of PolyIC and PD-1 mAb in unresectable late-stage HCC patients.

DETAILED DESCRIPTION:
Nowadays, primary liver cancer, especially hepatocellular carcinoma (HCC) has become the second leading cause of cancer-related death. Unfortunately, the therapeutic strategies are still limited for HCC. For HCC patients at advanced stage, up to now, sorafenib and regorafenib are applied for palliative therapy to prolong the patients' life. PD-1 blockade has became a promising immunotherapeutic strategy in many cancers. While it showed limited efficacy in liver cancer. Polyinosinic-polycytidylic acid (PolyIC) has been widely studied as a new anti-tumor drug and recent study showed that polyIC and PD-L1 mAb has a quite synergetic effect on the treatment of HCC. This study is aimed to evaluate the safety and efficacy of the combination of PolyIC and PD-1 mAb in unresectable late-stage HCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatocellular carcinoma with imaging diagnosis, in barcelona stage C, or stage B but resistant/recurrent to prior local treatment (e.g., TACE).
2. Eastern cooperative oncology group physical fitness score: 0-2.
3. Predicted survival time≥3 months.
4. Liver function of Child-Pugh A-B, no hepatic encephalopathy or physical examined ascites.
5. Routine blood tests were in accordance with the following criteria:

   White blood cell (WBC)≥2.0x10^9/L, Neutrophil≥1.0x10^9/L, platelet (PLT)≥50x10^9/L, hemoglobin (HB)≥80 g/dL, creatinine≤1.5xULN (upper limit of normal value), Alanine transaminase (ALT) and aspartate aminotransferase (AST)≤5xULN, total bilirubin (TB)≤51.3umol/L, international normalized ratio (INR) or prothrombin time (PT)≤1.7xULN, activated partial thromboplastin time (APTT)≤1.5xULN, serum albumin≥28g/L
6. Patients will be informed consent, and understand and are willing to cooperate with the trial and sign related documents.

Exclusion Criteria:

1. Has a history of malignant tumor in last 2 years, except basal and skin squamous cell carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma, superficial bladder cancer and carcinoma in situ of breast.
2. Received the treatment of polyIC or immune checkpoint inhibitors (e.g., PD-1/PD-L1 mAb or CTLA-4 mAb) in last 2 years.
3. Received the therapies of multi-kinase inhibitors (e.g., sorafenib, regorafenib), systemic chemotherapy, local therapy (e.g., TACE, radiotherapy), vaccination, immunomodulating therapy （e.g., interleukins, thymosin） or any other clinical trial in last 4 weeks.
4. Received any corticosterone or immunosuppressive drug in last 2 weeks.
5. Toxicity induced by previous anti-tumor therapies has not returned to the status of baseline or stability.
6. HIV positive (including previous anti-retroviral therapy), active HCV infection or active syphilis.
7. Any severe liver disease (e.g., severe liver cirrhosis, severe liver adenoma)
8. Any active or recurrent autoimmune disease.
9. Any interstitial pneumonia, non-infectious pneumonia, or uncontrolled systemic disease (e.g., uncontrolled hypertension or diabetes).
10. Severe cardiovascular risk factors.
11. Has a history of allogeneic stem cell transplantation or organ transplantation.
12. Imaging confirmed brain or meninges metastases.
13. Has the plan of pregnancy, or lactation.
14. Any kind of psychiatric disease or laboratory test abnormality that may result in the subject's failure to fully comply with the laboratory protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-10-22 (Estimated); Study Completion 2023-10-22 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 5 years
  Percentage of patients whose cancer shrinks or disappears after treatment

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 5 years
  Percentage of patients whose cancer doesn't progress after treatment
Progression free survival (PFS) | Up to approximately 5 years
  The percentage of people does not get worse for a period of time after diagnosis
Overall survival (OS) | Up to approximately 5 years
  The percentage of people still alive for a given period of time after diagnosis
Number of participants with treatment-related adverse events | Up to approximately 5 years
  Number of participants with treatment-related adverse events after drug initiation, as assessed by CTCAE v4.0
Percentage of participants with a better life quality | Up to approximately 5 years
  The percentage of participants with a better life quality after treatment, assessed by the questionnaires of European Organization for Research and Treatment of Cancer Quality of Life
Level of alpha-fetoprotein (AFP) | Up to approximately 5 years
  The percentage of participants with a decreased serum level of alpha-fetoprotein (AFP) after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, MD PhD, Principal Investigator — second affiliated hospital, Zhejiang University School of Medicine
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided